CLINICAL TRIAL: NCT00052780
Title: Phase I Trial of Temozolomide and O6-Benzylguanine in Pediatric Patients With Recurrent Brain Tumors
Brief Title: Temozolomide and O6-Benzylguanine in Treating Children With Recurrent Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03174; NCI-2012-03174 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR653709; PBTC-005 (Other: Pediatric Brain Tumor Consortium); PBTC-005 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Childhood Central Nervous System Germ Cell Tumor; Childhood Choroid Plexus Tumor; Childhood Craniopharyngioma; Childhood Ependymoblastoma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood High-grade Cerebellar Astrocytoma; Childhood High-grade Cerebral Astrocytoma; Childhood Infratentorial Ependymoma; Childhood Low-grade Cerebellar Astrocytoma; Childhood Low-grade Cerebral Astrocytoma; Childhood Medulloepithelioma; Childhood Mixed Glioma; Childhood Oligodendroglioma; Childhood Supratentorial Ependymoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway and Hypothalamic Glioma
MeSH Terms: conditions — Choroid Plexus Neoplasms; Astrocytoma; Oligodendroglioma; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma | interventions — O(6)-benzylguanine; Temozolomide; Filgrastim; Granulocyte Colony-Stimulating Factor

ARMS (1):
- Treatment (temozolomide, O6-benzylguanine) (Experimental): See Detailed Description
  Interventions: Drug: O6-benzylguanine; Drug: temozolomide; Biological: filgrastim; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: O6-benzylguanine — Given IV
  Other Names: BG
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Biological: filgrastim — Given SC or IV
  Other Names: G-CSF; Neupogen
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase I trial to study the safety of combining O6-benzylguanine with temozolomide in treating children who have recurrent or refractory brain tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. O6-benzylguanine may increase the effectiveness of temozolomide by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of temozolomide (Temodar) when administered with O6-benzylguanine (O6-BG) with and without G-CSF support to pediatric patients with refractory brain tumors stratified by previous radiotherapy.

SECONDARY OBJECTIVES:

I. To characterize the pharmacokinetics of temozolomide and O6-BG when used in combination.

II. To characterize toxicities associated with the combination of O6-BG and temozolomide with and without G-CSF support.

III. To document antitumor response in patients when treated with O6-BG and temozolomide.

IV. To determine the levels of MGMT enzyme and mismatch repair (MMR) proteins in tumor tissue, investigating a possible correlation with patient outcome.

OUTLINE: This is a dose-escalation study of temozolomide with and without filgrastim (G-CSF). Patients are stratified according to prior radiotherapy (RT)/myeloablative therapy (no RT or focal RT vs craniospinal RT or myeloablative therapy).

Patients receive O6-benzylguanine IV continuously on days 1 and 2 and oral temozolomide on day 1. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 2-6 patients in each stratum receive escalating doses of temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 25% of patients experience DLT. Once the MTD is determined, additional patients are treated at that dose level for a total of 12 patients treated at the MTD.

For courses 1-12, patients experiencing neutropenia may also receive G-CSF subcutaneously or IV daily beginning on day 3 and continuing until blood counts recover.

If neutropenia is the dose-limiting toxicity (DLT) for the first 2 strata, patients are further stratified according to concurrent G-CSF support (yes vs no).Cohorts of 3-6 patients in each stratum receive escalating doses of temozolomide with G-CSF until the MTD is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience DLT. Once the MTD is determined, 6 additional patients are treated at that dose.

Patients are followed for resolution of all adverse events occurring while on treatment and/or within 30 days of the last administration of study drug. Patients will be followed for the shortest of 1) three months after the last protocol based treatment, or 2) the date other therapy is initiated.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or refractory pediatric brain tumors; a histopathologic diagnosis from either the initial presentation or at the time of recurrence is required for all but brain stem gliomas
* Karnofsky or Lansky ≥ 60%
* Life expectancy > 8 weeks
* Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to study entry
* Chemotherapy: No more than 2 previous chemotherapy/biologic therapy regimens; evidence of recovery from prior chemotherapy/biologic therapy; no myelosuppressive chemotherapy within 3 weeks (6 weeks if a nitrosourea agent) of study entry; patients who have received temozolomide are eligible if they have not received the drug in the past 3 months and did not experience any non-hematopoietic Grade 3/4 toxicity with prior temozolomide therapy
* XRT: ≥ 3 months prior to study entry for craniospinal irradiation (≥ 18 Gy); ≥ 4 weeks for local radiation to primary tumor; and ≥ 2 weeks prior to study entry for focal irradiation to symptomatic metastatic sites
* Bone Marrow Transplant: ≥ 6 months prior to study entry
* Anti-convulsants: Patients will be eligible for this study even if they are receiving anti-convulsants
* Growth factors: Off all colony forming growth factor(s) > 2 weeks prior to study entry (G-CSF, GM-CSF, Erythropoietin)
* Dexamethasone: Patients who are receiving dexamethasone must be on a stable dose for at least 1 week prior to study entry
* ANC > 1,000/μl
* Platelets > 100,000/μl
* Hemoglobin > 8g/dl
* Patients may have bone marrow involvement by disease; platelet and Hgb counts must be transfusion independent
* Creatinine ≤ 1.5 times institutional normal for age
* Or GFR > 70 ml/min/1.73m^2
* Bilirubin ≤ upper limit of normal for age
* SGPT (ALT) < and SGOT (AST) < 2.5X institutional normal
* No overt renal, hepatic, cardiac or pulmonary disease
* Female patients of childbearing potential must have negative serum or urine pregnancy test; patient must not be pregnant or breast-feeding; while no known teratogenic effects are known for O6-BG so far, there is little data to address this specifically; as such, the prudent approach is to exclude pregnant and breastfeeding patients until further data is available
* Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study
* Signed informed consent according to institutional guidelines must be obtained and patients must begin therapy within seven (7) days of registration

Exclusion Criteria:

* Patients must not be receiving any other anticancer or experimental drug therapy
* Patients with a history of hypersensitivity to dacarbazine, temozolomide or polyethylene glycol are excluded

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2002-10; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
MTD of temozolomide | 28 days

SECONDARY OUTCOMES:
Pharmacokinetic parameters | Baseline and courses 1 and 3
  Summarized using descriptive statistics (mean, standard deviation) if normally distributed. For log-normally distributed data, the geometric mean will be used. If the data are not normally distributed, nonparametric statistics (median, minimum, maximum, interquartile ranges) will be used. Logistic regression models will be used to explore possible relationships between the systemic exposure to temozolomide, O6-benzylguanine, and their respective metabolites and toxicities and antitumor activity.
Acute toxicities | 4 weeks (course 1)
  These toxicities will be tabulated according to dose level.
Chronic toxicities | Up to 30 days post-treatment
  Tabulated according to dose level and course of therapy.
Histological response | Up to 5 years
  Exact confidence interval estimates of traditional response by histologic tumor type will be developed.
Duration of disease control | Up to 5 years
  Kaplan-Meier estimates will also be provided.
Survival | Up to 5 years
  Kaplan-Meier estimates will also be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (1):
- Pediatric Brain Tumor Consortium, Memphis, Tennessee, United States